CLINICAL TRIAL: NCT02004756
Title: Mechanisms of Dysfunction and the Influence of Exercise on Cardiac and Musculoskeletal Function in Children After the Fontan Procedure
Brief Title: Mechanisms of Dysfunction and the Influence of Exercise on Cardiac and Musculoskeletal Function
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Feasibility issues
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000016650
Record Dates: First submitted 2013-08-25; First posted 2013-12-09 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Congenital Heart Disease
Keywords: pediatric; fontan; congenital heart disease; cardiac and musculoskeletal funion; cardiac and/or musculoskeletal metabolism; exercise training intervention
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fontan Patients (Experimental): Fontan patients who are monitored at the Hospital for Sick Children (SickKids) will undergo an exercise program
  Interventions: Other: Exercise Program
- Healthy Controls (No Intervention): Healthy age-matched adolescents

INTERVENTIONS:
Other: Exercise Program — The Fontan cohort will subsequently complete a 12-week moderate intensity exercise intervention whereby individualized activity-based home interventions will be prescribed (i.e., sample activities: walking, jogging, swimming, cycling, soccer). More specifically, individualized weekly exercise programs for participants will be provided incorporating two specific exercise components.
  Arms: Fontan Patients

SUMMARY:
Primary Objective: To determine if impairments in cardiac and musculoskeletal function and metabolism exist in Fontan children.

Secondary Objectives:

1. To determine if impairments do exist, are they related to exercise capacity.
2. To determine if a 12-week exercise training intervention improves cardiac and/or musculoskeletal metabolism.

Hypothesis: The investigators hypothesize that abnormalities in cardiac and skeletal function are evident, influence exercise capacity, and can be improved with exercise training.

DETAILED DESCRIPTION:
This proposed research provides an interdisciplinary approach to understanding exercise intolerance by examining cardiac and musculoskeletal metabolism in a unique cohort of children with congenital heart disease. Study findings may more importantly lead to evidence-based exercise interventions that promote improvements in overall physical health, quality of life, and functional status for Fontan children. Furthermore, this pilot study will lead to the development of a novel research protocol which may be applied to larger Fontan and other congenital heart disease cohorts. This study will also provide preliminary data to develop and conduct a larger clinical research project.

ELIGIBILITY:
Inclusion Criteria:

Fontan Patients:

1. Patients who have had the Fontan cardiac procedure
2. 10-16 years of age
3. Written Informed Consent

Healthy Controls:

1. 10 - 16 years of age
2. Written Informed Consent

Exclusion Criteria:

Fontan Patients:

1. Contraindication to exercise
2. Physically active (i.e., ≥ 60 minute of moderate-vigorous activity) (Strong et al., 2005)
3. Patients in whom MRI is contraindicated (e.g. pacemaker, ocular metal, claustrophobia, tattoos)
4. Patients with a known allergy to gadolinium.
5. Patients with a history of allergic disposition or have anaphylactic reactions
6. Moderate-to-severe renal impairment (defined as having a GFR/ eGFR < 60 mL/min)
7. Have Sickle Cell anemia
8. Known pregnancy, or breast feeding
9. Patient is uncooperative during a MRI without sedation or anesthesia

Healthy Controls:

1. Contraindication to exercise
2. Physically active (i.e., ≥ 60 minute of moderate-vigorous activity) (Strong et al., 2005)
3. Patients in whom MRI is contraindicated (e.g. pacemaker, ocular metal, claustrophobia, tattoos, pregnancy)
4. Patient is uncooperative during a MRI without sedation or anesthesia

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Cardiac and skeletal function and metabolism | 1 day
  Blood oxygen level dependent functional magnetic resonance imaging (BOLD fMRI), and 31P-MRS will allow for the precise measurement of cardiac and musculoskeletal function, circulatory perfusion and vascular reactivity, and aerobic and anaerobic metabolism, respectively. Cardiac function will be examined via MRI and exercise echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Brian McCrindle, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada